CLINICAL TRIAL: NCT00488228
Title: Behavioral Self-Regulation for Weight Loss in Young Adults
Brief Title: Behavioral Self-Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMTT# 2096-07
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2008-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Professional Autonomy

ARMS (2):
- 1 (Experimental): Participants in the behavioral self-regulation intervention will receive a modified standard treatment that incorporates daily weighing and training in self-regulation methods for weight loss. All treatment modules are adapted for a young adult age group.
  Interventions: Behavioral: self-regulation
- 2 (Experimental): Participants in the Standard group will receive a brief version of standard behavioral weight loss treatment with treatment modules tailored to better meet the needs of young adults.
  Interventions: Behavioral: self-regulation

INTERVENTIONS:
Behavioral: self-regulation — The current study involves a behavioral weight loss intervention tailored specifically to young adults. All participants receive calorie and activity prescriptions as well as training in behavior modification. In addition, one group receives training in self-regulation techniques using daily weighing.

SUMMARY:
The purpose of this pilot study is to determine whether incorporating self-regulation training using daily weighing is efficacious within a behavioral weight loss program specifically targeting young adults.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 27 and 40
* age between 21 and 35

Exclusion Criteria:

* report a history of eating disorder or a current eating disorder
* report a heart condition or other medical condition that would limit ability to participate in an exercise program without direct supervision from physician
* report major psychiatric diseases or organic brain syndromes
* currently participating in another weight loss program, are taking a weight loss medication, or have lost more than 5% of body weight curing last 6 months
* pregnant, lactating, or less than 6 months post-partum
* intend to move out of city within the time frame of the investigation or will miss multiple meetings during the study time frame

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
weight change | 10 weeks and 20 weeks

SECONDARY OUTCOMES:
eating disorder symptoms, physical activity, body image, mood symptoms, and self-efficacy about eating behavior | 10 weeks and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G LaRose, Ph.D., Study Director — The Miriam Hospital; Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Gokee-Larose J, Gorin AA, Wing RR. Behavioral self-regulation for weight loss in young adults: a randomized controlled trial. Int J Behav Nutr Phys Act. 2009 Feb 16;6:10. doi: 10.1186/1479-5868-6-10. PMID 19220909